CLINICAL TRIAL: NCT02865109
Title: Expanded Access Program (EAP) to Provide Nusinersen to Patients With Infantile-onset Spinal Muscular Atrophy (SMA)
Brief Title: Expanded Access Program (EAP) for Nusinersen in Participants With Infantile-onset (Consistent With Type 1) Spinal Muscular Atrophy (SMA)
Status: No longer available | Type: Expanded Access
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 232-SM-901
Record Dates: First submitted 2016-08-10; First posted 2016-08-12 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Infantile-onset Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; SMA; SMN; SMNRx; ISIS-SMNRx; ISIS-SMN Rx; ISIS 396443; ISIS-396443; ENDEAR; IONIS-SMNRx; IONIS-SMN Rx; EMBRACE; NURTURE; IONIS; BIOGEN; SHINE; Nusinersen
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Nusinersen — Administered by intrathecal injection
  Other Names: ISIS 396443; BIIB058; Spinraza

SUMMARY:
To provide access to nusinersen to eligible patients with Infantile-onset Spinal Muscular Atrophy (SMA) (consistent with Type 1) to address a high-unmet medical need.

DETAILED DESCRIPTION:
The nusinersen expanded access program (EAP) is available at approved treatment centers in select territories.

A doctor must decide whether nusinersen treatment is appropriate for each patient, based on the patient's medical history and program eligibility criteria. A full list of participating treatment centers is provided in the 'Contacts and Locations' section of this listing, and is regularly updated.

Following local approval and official reimbursement of nusinersen in each territory, the EAP will close and patients will transfer to commercially available drug.

ELIGIBILITY:
Key Inclusion Criteria:

* Genetic documentation of 5q SMA homozygous gene deletion, homozygous mutation, or compound heterozygote.
* Onset of clinical signs and symptoms at ≤ 6 months (180 days) of age, consistent with infantile onset, Type I SMA
* Patient whose care in the opinion of the treating physician meets, and is expected to continue to meet, the guidelines set out in the 2007 Consensus Statement for Standard of Care in SMA

Key Exclusion Criteria:

* Patient is qualified to participate in an ongoing clinical trial with nusinersen
* Participation in a prior nusinersen study
* Previous exposure to nusinersen
* History of brain or spinal cord disease that would interfere with the LP procedures or CSF circulation
* Presence of implanted shunt for the drainage of CSF or implanted CNS catheter
* Previous or current participation in a clinical trial with an investigational gene therapy for SMA
* Participation in a study with an investigational therapy for SMA within 6 months or five half-lives of the investigational drug, whichever is the longer, prior to the first dose of nusinersen.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (7):
- Hospital Pablo Tobon Uribe, Medellín, Colombia
- New Zealand (2):
  - Auckland City Hospital, Grafton, Auckland
  - Auckland District Health Board ADHB, Grafton, Auckland
- Turkey (Türkiye) (4):
  - Erciyes University Hospital, Kayseri, Anatolia
  - Hacettepe University, Ankara, Central Anatolia
  - Marmara Uni. Research & Educational Hospital, Kadıköy, Istanbul
  - Medipol University Hospital, Istanbul, Marmara